CLINICAL TRIAL: NCT04864171
Title: REvelation of PAthophySiological PhenotypeS of VUlneRable Lipid-Rich PlaquE on Near-InfraRed Spectroscopy: REASSURE-NIRS
Brief Title: REASSURE-NIRS Registry
Acronym: REASSURENIRS
Status: Recruiting | Type: Observational
Sponsor: National Cerebral and Cardiovascular Center, Japan (Other)
Responsible Party: Principal Investigator, Yu Kataoka, Chief consultant, National Cerebral and Cardiovascular Center, Japan
Other Study IDs: M30-084-4
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lipid-Rich Atherosclerosis of Coronary Artery
Keywords: near-infrared spectroscopy; lipid-rich plaque; coronary artery disease; intravascular imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: near-infrared spectroscopy — Near-infrared spectroscopy is an intravascular imaging device to visualize lipid-rich plaque of coronary artery.

SUMMARY:
RESSURE-NIRS registry is designed to investigate clinical and pathophysiological characteristics of NIRS-derived lipid-rich plaque in patients with coronary artery disease. This is an on-going multi-center prospective registry in Japan.

DETAILED DESCRIPTION:
NIRS imaging is an invasive intravascular imaging modality to quantitatively visualize lipid-rich atheroma in vivo. While NIRS-derived lipid-rich plaque has been shown to associate with cardiovascular events, there is limited clinical data about the association of this high-risk plaque with risk factors, medication use, prognosis and response of PCI. RESSURE-NIRS registry is an on-going multi-center prospective registry in Japan, which enroll subjects with coronary artery disease who received NIRS imaging to evaluate coronary atherosclerosis. The primary outcome is maximum 4-mm lipid core burden index at coronary lesions measured by NIRS imaging. Secondary major outcomes include entire lipid core burden index, plaque volume, plaque attenuation and echo-lucent area. The anticipated number of study subjects is 2000 cases.

ELIGIBILITY:
Inclusion Criteria:

patients with coronary artery disease clinical indication for coronary angiography and/or percutaneous coronary intervention visualization of coronary lesions with NIRS

Exclusion Criteria:

poor quality of NIRS images

Ages: 20 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population should be patients with coronary artery disease who requires coronary angiography and/or percutaneous coronary intervention with NIRS imaging
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
MACE | at an average of 3 year
  major adverse cardiovascular events (=cardiac-cause death, non-fatal MI and clinically-driven non-restenotic coronary revascularization)

SECONDARY OUTCOMES:
Coronary physiological characteristics at lipid-rich plaques | Physiological measures are collected during the procedure: percutaneous coronary intervention
  Identify and quantify coronary physiological findings (=fractional flow reserve and delta fractional flow reserve) for cardiovascular risk stratification of persons with lipid-rich plaques.

OTHER OUTCOMES:
The occurrence of MACE in patients who achieved LDL-C <1.4 mmol/L | at an average of 2 year
  The efficacy of LDL-C <1.4 mmol/L on MACE
gender difference in NIRS-derived measures | NIRS-derived measures are collected during the procedure
  sex-related difference in maxLCBI

CONTACTS AND LOCATIONS:
Overall Officials: Yu Kataoka, MD, Principal Investigator — National Cerebral & Cardiovascular Center
Locations (2):
- Japan (2):
  - Miyazaki Medical Association Hospital, Miyazaki
  - National Cerebral & Cardiovascular Center, Suita

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kataoka Y, Puri R, Andrews J, Honda S, Nishihira K, Asaumi Y, Noguchi T, Yasuda S, Nicholls SJ. In vivo visualization of lipid coronary atheroma with intravascular near-infrared spectroscopy. Expert Rev Cardiovasc Ther. 2017 Oct;15(10):775-785. doi: 10.1080/14779072.2017.1367287. Epub 2017 Aug 28. PMID 28846060
- [Background] Kitahara S, Kataoka Y, Miura H, Nishii T, Nishimura K, Murai K, Iwai T, Nakamura H, Hosoda H, Matama H, Doi T, Nakashima T, Honda S, Fujino M, Nakao K, Yoneda S, Nishihira K, Kanaya T, Otsuka F, Asaumi Y, Tsujita K, Noguchi T, Yasuda S. The feasibility and limitation of coronary computed tomographic angiography imaging to identify coronary lipid-rich atheroma in vivo: Findings from near-infrared spectroscopy analysis. Atherosclerosis. 2021 Apr;322:1-7. doi: 10.1016/j.atherosclerosis.2021.02.019. Epub 2021 Feb 24. PMID 33706078
- [Background] Imamoto K, Kataoka Y, Hosoda H, Noguchi T. Suboptimal lipoprotein (a) control and residual plaque instability despite proprotein convertase subtilisin/kexin type 9 inhibitor use in heterozygous familial hypercholesterolaemia: insights from serial near-infrared spectroscopy imaging. Eur Heart J. 2021 Jun 7;42(22):2218-2219. doi: 10.1093/eurheartj/ehab218. No abstract available. PMID 33822931
- [Background] Puri R, Madder RD, Madden SP, Sum ST, Wolski K, Muller JE, Andrews J, King KL, Kataoka Y, Uno K, Kapadia SR, Tuzcu EM, Nissen SE, Virmani R, Maehara A, Mintz GS, Nicholls SJ. Near-Infrared Spectroscopy Enhances Intravascular Ultrasound Assessment of Vulnerable Coronary Plaque: A Combined Pathological and In Vivo Study. Arterioscler Thromb Vasc Biol. 2015 Nov;35(11):2423-31. doi: 10.1161/ATVBAHA.115.306118. Epub 2015 Sep 3. PMID 26338299
- [Background] Kitahara S, Kataoka Y, Sugane H, Otsuka F, Asaumi Y, Noguchi T, Yasuda S. In vivo imaging of vulnerable plaque with intravascular modalities: its advantages and limitations. Cardiovasc Diagn Ther. 2020 Oct;10(5):1461-1479. doi: 10.21037/cdt-20-238. PMID 33224768
- [Background] Hosoda H, Kataoka Y, Otsuka F, Yasuda S. Severely calcified lipidic atheroma on intravascular ultrasound and near-infrared spectroscopy imaging: its association with slow-flow phenomenon during percutaneous coronary intervention. Eur Heart J Case Rep. 2019 Jun 1;3(2):ytz078. doi: 10.1093/ehjcr/ytz078. No abstract available. PMID 31449658
- [Background] Nishihira K, Yamashita A, Kataoka Y, Shibata Y, Asada Y. Visualization of oxidized low-density lipoprotein at lipid-rich plaque in a ST-segment elevation myocardial infarction case with heterozygous familial hypercholesterolaemia: insights from near-infrared spectroscopy and histopathological analysis. Eur Heart J Cardiovasc Imaging. 2019 Nov 1;20(11):1316. doi: 10.1093/ehjci/jez156. No abstract available. PMID 31180473
- [Background] Kaichi R, Kataoka Y, Yasuda S. Erupted coronary atheroma: insights from multi-modality imaging. Int J Cardiovasc Imaging. 2018 Oct;34(10):1669-1671. doi: 10.1007/s10554-018-1378-1. Epub 2018 May 24. PMID 29799063
- [Background] Nishihira K, Otsuka F, Kataoka Y, Asaumi Y, Kaneta K, Nakano H, Ohta-Ogo K, Ishibashi-Ueda H, Noguchi T, Yasuda S. Embolization of Neoatherosclerosis After Percutaneous Coronary Intervention: Insights From Near-Infrared Spectroscopy Imaging and Histopathological Analysis. Circ Cardiovasc Interv. 2018 Feb;11(2):e006175. doi: 10.1161/CIRCINTERVENTIONS.117.006175. No abstract available. PMID 29445002
- [Background] Nishihira K, Asaumi Y, Kataoka Y, Ishibashi-Ueda H, Yasuda S. In vivo comparison of lipid-rich plaque on near-infrared spectroscopy with histopathological analysis of coronary atherectomy specimens. Eur Heart J Cardiovasc Imaging. 2018 Jan 1;19(1):116. doi: 10.1093/ehjci/jex247. No abstract available. PMID 29040461
- [Derived] Gilard M, Wijns W. High-Intensity Lipid-Lowering Therapies: An Opportunity for Improving Cardiovascular Outcomes in Postmenopausal Women? Circ Cardiovasc Imaging. 2023 May;16(5):e015544. doi: 10.1161/CIRCIMAGING.123.015544. Epub 2023 May 10. No abstract available. PMID 37161823
- [Derived] Kataoka Y, Nicholls SJ, Puri R, Kitahara S, Kiyoshige E, Nishimura K, Murai K, Iwai T, Sawada K, Matama H, Honda S, Takagi K, Fujino M, Yoneda S, Otsuka F, Nishihira K, Takamisawa I, Asaumi Y, Noguchi T. Sex Differences in the Density of Lipidic Plaque Materials: Insights From the REASSURE-NIRS MultiCenter Registry. Circ Cardiovasc Imaging. 2023 May;16(5):e015107. doi: 10.1161/CIRCIMAGING.122.015107. Epub 2023 May 10. PMID 37161775
- [Derived] Nakamura H, Kataoka Y, Nicholls SJ, Puri R, Kitahara S, Murai K, Sawada K, Matama H, Iwai T, Honda S, Fujino M, Takagi K, Yoneda S, Otsuka F, Nishihira K, Asaumi Y, Tsujita K, Noguchi T. Elevated Lipoprotein(a) as a potential residual risk factor associated with lipid-rich coronary atheroma in patients with type 2 diabetes and coronary artery disease on statin treatment: Insights from the REASSURE-NIRS registry. Atherosclerosis. 2022 May;349:183-189. doi: 10.1016/j.atherosclerosis.2022.03.033. Epub 2022 Apr 10. PMID 35450750